CLINICAL TRIAL: NCT03022383
Title: TopQ Cutoff Threshold Validation Study for DRI OCT Triton Plus
Status: Completed | Type: Observational
Sponsor: Topcon Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Organization: Topcon Corporation (Industry)
Other Study IDs: Topcon Triton 1222-2016
Record Dates: First submitted 2017-01-11; First posted 2017-01-16 (Estimated); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Healthy Eyes
Keywords: no known ocular pathology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects Presenting With Normal Eyes: Subjects with no known ocular diseases will be scanned on the DRI OCT Triton Plus device
  Interventions: Device: DRI OCT Triton plus

INTERVENTIONS:
Device: DRI OCT Triton plus — OCT Machine used for diagnostic purposes

SUMMARY:
To determine optimal cut-off value for the TopQ cut-off on the DRI OCT Triton plus

DETAILED DESCRIPTION:
Scans with a TopQ score below the optimum cut-off should be considered to be poor or unacceptable quality, and scans with a TopQ score above the cut-off should be considered good or acceptable quality. The study will evaluate the predetermined cut-off values by investigating measurement variability of scans.

ELIGIBILITY:
Inclusion Criteria

* Participants must be at least 18 years of age
* Participants must be able to complete all testing (all OCT scans)
* Participants must volunteer to be in the study and sign the consent form

Exclusion Criteria

* Subject with history of ocular disease or ocular pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with no known eye disease.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-01; Primary Completion 2017-02 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Measurement Variability of Signal to Noise Ratio | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Chieh Huang, PhD, Principal Investigator — Topcon Medical Systems, Inc.
Locations (1):
- Topcon Medical Systems Inc., Oakland, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided